CLINICAL TRIAL: NCT00329745
Title: A Phase III, Double-blind, Randomized, Placebo-controlled, Multi-country and Multi-center Study to Assess the Efficacy and Safety of Two Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants.
Brief Title: Year 3 Extension for Efficacy Follow-up in Subjects Vaccinated in Studies Rota-028, 029 or 030 (NCT00197210)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 107070; 107072 (Other: GSK); 107076 (Other: GSK); NCT00329953 (obsolete NCT alias); NCT00331734 (obsolete NCT alias)
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Results first posted 2009-10-14 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Infections, Rotavirus
Keywords: Rotavirus Gastroenteritis; Human rotavirus vaccine, efficacy, infants
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Rotarix Group (Experimental): During the primary study (NCT00197210) subjects received two oral doses of Rotarix™ vaccine.
  Interventions: Biological: Rotarix™
- Placebo Group (Placebo Comparator): During the primary study (NCT00197210) subjects received two oral doses of placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Rotarix™ — Oral administration, 2 doses
  Arms: Rotarix Group
Biological: Placebo — Oral administration, 2 doses
  Arms: Placebo Group

SUMMARY:
This Year 3 extension of the main study rota-028, 029 or 030 is conducted to evaluate vaccine efficacy against severe rotavirus (RV) gastroenteritis (GE) during third year of life in infants previously vaccinated with human rotavirus (HRV) vaccine or placebo in the following schedules:

at 3 and 4 months of age in study rota-028; at 2 and 4 months of age in study rota-029 or rota-030.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Note that no new subjects will be recruited in this extension phase studies.

The expected total enrolment for the primary studies was as follows:

rota-028: 5700 rota-029: 3018 rota-030: 1102

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including, 6 and 12 weeks of age in Hong Kong and Taiwan or 11 to 17 weeks of age in Singapore at the time of the first vaccination according to the country recommendations for the routine vaccination schedules.
* Written informed consent obtained from the parent or guardian of the subject, prior any study procedure.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine or placebo, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* Child is unlikely to remain in the study area for the duration of the study
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period. Oral intake of immunoglobulins is allowed.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal tract or other serious medical condition as determined by the investigator.
* First or second degree of consanguinity of parents.

Ages: 2 Years to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8687 (Actual)
Dates: Start 2007-01; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Reference to the Primary Study NCT number — http://www.clinicaltrials.gov/ct/show/NCT00197210
- Available data/document: Informed Consent Form: 107070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register. The results of this study 107070 are summarised with studies 444563/028, 444563/029, 444563/030, 107072, and 107076 on the GSK Clinical Study Register.
- Available data/document: Statistical Analysis Plan: 107070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107070 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 4359 | 4328
Completed | 4272 | 4226
Not Completed | 87 | 102
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 86 | 101

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 4359 | 4328 | 8687
Age, Continuous [Mean (Standard Deviation); unit: months] | 35.4 (1.18) | 35.4 (1.26) | 35.4 (1.22)
Gender [Count of Participants; unit: Participants]
  Female | 2108 | 2097 | 4205
  Male | 2251 | 2231 | 4482

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Severe Rotavirus Gastroenteritis (RV GE) Caused by the Circulating Wild-type Rotavirus Strains
Description: Severe RV GE is an episode of severe GE in which rotavirus other than vaccine strain was identified in a GE stool sample.
  Note that this outcome measure is secondary in the study protocol. We have reported it here as primary outcome measure, since none of the primary outcome measures in the study protocol pertain to the time point (Year 3 follow-up) presented in this summary.
Time Frame: From Year 2 up to Year 3
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for efficacy.
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 4222 | 4185
subjects | 0 | 13

2. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: An SAE is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: From the end of the primary study up to Year 3
Measure: Number; unit: subjects
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 4359 | 4328
subjects | 10 | 11

ADVERSE EVENTS:
Description: Adverse events were not systematically followed up in this study. Only the adverse events (and serious adverse events) leading to subject withdrawal or drop-out were collected.
Arm/Group | Rotarix Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 10/4359 | 11/4328
Other Adverse Events (participants affected / at risk) | 0/4359 | 0/4328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=4359) | Placebo Group (N=4328)
Gastroenteritis (Infections and infestations) | 3 | 2
Intussusception (Gastrointestinal disorders) | 2 | 1
Upper respiratory tract (Infections and infestations) | 0 | 3
Gastritis (Gastrointestinal disorders) | 1 | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 1
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Croup infectious (Injury, poisoning and procedural complications) | 0 | 1
Dehydratation (Metabolism and nutrition disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Epyema (Infections and infestations) | 0 | 1
Febrile convulsion (Nervous system disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Kawasaki's disease (Infections and infestations) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.